CLINICAL TRIAL: NCT04623229
Title: A Comparison of Patient Perceptions Undergoing Manual Cataract Surgery (MCS) vs Refractive Laser-assisted Cataract Surgery (ReLACS) in First and Second Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UptownEye
Record Dates: First submitted 2020-07-09; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: MCS vs ReLACS; Pain Perception Postoperatively First Eye vs Second Eye; Early Anesthesia vs Standard Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MCS (Experimental)
  Interventions: Procedure: MCS
- ReLACS Early (Experimental)
  Interventions: Procedure: ReLACS Early
- ReLACS Standard (Experimental)
  Interventions: Procedure: ReLACS Standard

INTERVENTIONS:
Procedure: MCS — Manual Cataract Surgery
  Arms: MCS
Procedure: ReLACS Early — ReLACS with early administration of anesthesia
  Arms: ReLACS Early
Procedure: ReLACS Standard — ReLACS with standard time administration of anesthesia
  Arms: ReLACS Standard

SUMMARY:
The focus of this study is to assess how pain can be mitigated for patients undergoing cataract surgery through the early application of anesthesia prior to the surgery as compared to the standard timing, and by using the ReLACS cataract surgery technique compared to the standard MCS technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing uncomplicated cataract surgery with either surgical technique (MCS or ReLACS)
2. Patients who require surgery in both eyes by same surgeon
3. Able to understand English and complete a pain assessment

Exclusion Criteria:

1. Deafness or communication disorder, known Dementia, Severe COPD/Asthma (severe lung disorder), Severe OSA, Psychiatric or Anxiety conditions, involuntary movement disorders, allergy to the anesthesia, any conditions requiring intraoperative iris manipulation, any prior ocular surgery
2. Pre-existing chronic eye pain or uveitis, or complicated cataracts (dislocation, zonulopathy)
3. Pre-existing uncontrolled glaucoma/high IOP
4. Intraoperative complications or non-routine cataracts (eg. Sutures, excessive time of surgery)
5. Any patient who requires Deep Sedation (Propofol), GA or preOP Ativan
6. Patients under 40, severe obesity (BMI >35)
7. Chronic pain/narcotics/Recreational/medical marijuana

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Pain Perception between Manual Cataract Surgery and Refractive Laser Assisted Cataract Surgery | 1 year
  The pain scores will be measured using the Visual Analogue Scale (VAS) which is based on a 0 to 10 scale.

SECONDARY OUTCOMES:
Effects of Early vs Standard administration of neurolept anesthesia on pain perception | 1 year
  The pain scores will be measured using the Visual Analogue Scale (VAS) which is based on a 0 to 10 scale.
Differences in pain perception between first eye vs second eye | 1 year
  The pain scores will be measured using the Visual Analogue Scale (VAS) which is based on a 0 to 10 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Uptown Eye Speicialists, Brampton, Otario, Canada

IPD SHARING:
Plan to Share IPD: No